CLINICAL TRIAL: NCT04614363
Title: Comparison of 68 Ga-PSMA Positron Emission Tomography (PET)/CT to Conventional Imaging in Men With High Risk Prostate Cancer
Brief Title: 68 Ga-PSMA for High Risk Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Brian Miles, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00026240
Record Dates: First submitted 2020-10-08; First posted 2020-11-04 (Actual); Results first posted 2022-12-29 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer; High Risk
Keywords: PSMA; 68 Ga
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Intervention Model Description: All subjects will receive the Investigational Product.
Masking Description: To minimize bias, all PET/CT images will be interpreted by a board certified radiologist. They will be blinded to the final outcome, such as histopathology of any biopsies and the outcome of subsequent imaging.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68 Ga PSMA (Experimental): Comparison between the results of 68 Ga-PSMA PET/CT to conventional imaging (bone scan, CT) in men with high risk prostate cancer.
  Interventions: Drug: 68Ga-PSMA

INTERVENTIONS:
Drug: 68Ga-PSMA — All subjects enrolled in the study will receive a single IV dose of 3-7 mCi of 68 Ga-PSMA (study drug) followed by PET/CT imaging for detection of tumor location.
  Other Names: 68 Ga-PSMA 11

SUMMARY:
This is a prospective, single-center, open-label pilot study of 68GA-PSMA-11 given at a single time prior to PET/CT imaging in men with localized high risk prostate cancer or biochemical recurrence. The imaging agent (68 Ga-PSMA 11 will be administered on an outpatient basis. It will be administered prior to the PET/CT imaging. The objective is to evaluate the distribution of 68GA-PSMA-11 in tissues and to determine if this alters the planned clinical management.

DETAILED DESCRIPTION:
This is a prospective, open label, single-center, single-arm, pilot diagnostic accuracy study to evaluate the tissue distribution of 68Ga-PSMA Positron Emission Tomography (PET)/CT in 80 patients with high risk localized prostate cancer or biochemical recurrence.

Subjects will receive a single IV dose of 3-7 mCi of 68Ga-PSMA (study drug) followed by PET/CT imaging 60-90 minutes after injection. All patients will be closely monitored with vital signs (blood pressure and heart rate), before and 2 hours following radiotracer administration.

Patients will receive a phone call 2 days following PET/CT to assess for adverse events.

To minimize bias, all PET/CT images will be interpreted by a board-certified radiologist. The radiologist evaluating the images will be blinded to the final outcome, such as the histopathology of any biopsies and the outcome of subsequent imaging.

Patients with study-defined high-risk features who are eligible and scheduled for radical prostatectomy will undergo 68Ga-PSMA-11 PET/CT injection. The results of the 68Ga-PSMA-11 PET/CT may alter patient management in one of several ways, including the decision to not pursue surgical extirpation (e.g. in the event of extensive distant metastasis) in favor of systemic therapy. It is also possible that the extent of surgical resection may be altered, such as non-regional pelvic or retroperitoneal lymph node dissection. The alteration in planned surgical treatment from standard of care will be recorded as a secondary-end point.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 21 years or older
* Ability to understand and provide written informed consent
* All patients must have histopathological proven adenocarcinoma of the prostate
* ECOG performance status 0-1
* No evidence of other malignancy (except squamous or basal cell skin cancers)
* Consent to use acceptable form of birth control following the imaging period (condoms for a period of seven days after injection if sexually active)

A. Inclusion criteria specific for the pre-prostatectomy group:

Untreated prostate Cancer with high-risk features, as defined as having at least one of the following criteria:

i. PSA ≥ 20.0 ng/mL ii. ISUP Gleason Grade Group 3, 4 or 5 iii. Clinical stage T3

B. Inclusion criteria specific for biochemical recurrence:

(i) Histopathological proven prostate adenocarcinoma (ii)Rising PSA after definitive therapy with prostatectomy or radiation (therapy (external beam or brachytherapy).

1. Post radical prostatectomy (RP), PSA greater than or equal to 0.2 ng/ml measured more than 6 weeks after RP.
2. Post-radiation therapy, PSA that is equal to or greater than 2 ng/ml rise above PSA nadir

Exclusion Criteria:

* Unable to tolerate a PET/CT (e.g. unable to lie flat)
* Recent history of a secondary malignancy in the past year, excluding non-melanoma skin cancer (non-metastatic)
* Known allergic reactions to 68-Ga, or gadolinium-based contrast agents.
* Treatment with another investigational drug or other intervention 2 years.
* Patient has any medical, psychological or social condition that, in opinion of the investigator will make difficult for the participant to tolerate study intervention.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Miles, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Localized High Risk Prostate Cancer: Patients with high risk prostate cancer scheduled for prostatectomy will receive a single IV dose of 3-7 mCi of 68Ga-PSMA (study drug) followed by PET/CT imaging 60-90 minutes after injection.
- Biochemical Recurrence: Patients with biochemical recurrence post radical prostatectomy will receive a single IV dose of 3-7 mCi of 68Ga-PSMA (study drug) followed by PET/CT imaging 60-90 minutes after injection.
Period: Overall Study
Arm/Group | Localized High Risk Prostate Cancer | Biochemical Recurrence
Started | 30 | 50
Completed | 27 | 49
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: Patients with high risk prostate cancer scheduled for prostatectomy and patients with biochemical recurrence will receive a single IV dose of 3-7 mCi of 68Ga-PSMA (study drug) followed by PET/CT imaging 60-90 minutes after injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Localized High Risk Prostate Cancer | Biochemical Recurrence | Total
Number analyzed (Participants) | 30 | 50 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 19 | 33
  >=65 years | 16 | 31 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 50 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 27 | 45 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 22 | 48 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 50 | 80

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Lymph Node Involvement
Description: Number of patients with cTxNoMo (clinically localized disease) found on final histological examination to have lymph node involvement as determined by 68GA-PSMA-11 PET/CT.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Localized High Risk Prostate Cancer | Biochemical Recurrence
Number analyzed (Participants) | 30 | 50
Participants | 4 | 28

2. Primary Outcome: Proportion of Patients Which Clinical Management Was Altered
Description: Number of patients in which 68GA-PSMA-11 PET/CT altered the planned clinical management.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Groups:
- Biochemical Recurrence: Patients with biochemical recurrence will receive a single IV dose of 3-7 mCi of 68Ga-PSMA (study drug) followed by PET/CT imaging 60-90 minutes after injection.
Arm/Group | Localized High Risk Prostate Cancer | Biochemical Recurrence
Number analyzed (Participants) | 30 | 50
Participants | 2 | 30

3. Secondary Outcome: Intensity of Uptake as a Predictor of Clinical Outcome or Aggressiveness
Description: Uptake intensity detected on PET/CT in the prostate and outside of the prostate
Time Frame: 18 months
Measure: Mean (Full Range); unit: SUV
Arm/Group | Localized High Risk Prostate Cancer | Biochemical Recurrence
Number analyzed (Participants) | 30 | 50
SUV
  SUV (mean) inside the prostate : mean SUV | 22.45 [3.9 to 105.7] | 0 [0 to 0]
  SUV (mean) outside the prostate | 43.8 [12.8 to 74.9] | 16.9 [2.1 to 99.7]

4. Secondary Outcome: Number of Patients With Suspicious Lesions
Description: Number of patients in which 68Ga-PSMA 11 PET/CT showed suspicious lesions that are were not seen in standard diagnostic modalities of bone scan, CTs or MRI.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Localized High Risk Prostate Cancer | Biochemical Recurrence
Number analyzed (Participants) | 30 | 50
Participants | 4 | 17

ADVERSE EVENTS:
Time Frame: Participants were followed at 2 and 6 months post PET scan.
Groups:
- Localized High Risk Prostate Cancer: One patient was hospitalized due to acute CVA, grade 2, not related.
- Biochemical Recurrence: Two patients in this group died. These events were not related to the study. Acute encephalopathy and metastatic prostate cancer to liver, bone and brain.
Arm/Group | Localized High Risk Prostate Cancer | Biochemical Recurrence
All-Cause Mortality (participants affected / at risk) | 0/30 | 2/50
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/50
Other Adverse Events (participants affected / at risk) | 0/30 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Localized High Risk Prostate Cancer (N=30) | Biochemical Recurrence (N=50)
Encephalopathy (Nervous system disorders) | 0 | 1 (1) — Acute Encephalopathy, Grade 5, unrelated to study.
Prostate cancer metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) — Metastasis to liver, bone and brain, grade 5, unrelated to study.
Acute cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 — Acute CVA, grade 2, required hospitalization, unrelated to study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT04614363/Prot_SAP_000.pdf